CLINICAL TRIAL: NCT05022940
Title: Functional Evolution of Traumatic Brain Injured Adults During Rehabilitation and Social Participation: a Continuum of Care to Community Study
Brief Title: Functional Evolution of Traumatic Brain Injured Adults During Rehabilitation and Social Participation
Status: Recruiting | Type: Observational
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Michelle McKerral, Professor and Researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Other Study IDs: CRIR MMcK 2
Record Dates: First submitted 2021-08-17; First posted 2021-08-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Brain Injury
Keywords: Social participation; Quality of life
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Whole-Body Irradiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TBI rehabilitation: All individuals with mild, moderate or severe TBI registered into rehabilitation.
  Interventions: Other: Usual gold-standard multidisciplinary rehabilitation for TBI

INTERVENTIONS:
Other: Usual gold-standard multidisciplinary rehabilitation for TBI — In individual and group interventions within a holistic interdisciplinary rehabilitation program focusing on resumption of daily activities and social roles. Interventions could include physiotherapy or physical training, occupational therapy, speech therapy, and neuropsychology/psychology, which aimed at reducing the impacts of cognitive difficulties in daily life by using self-guided and environmental strategies.

SUMMARY:
The research project aims to better understand the multiple factors related to the clinical evolution and the social participation of traumatic brain injured (TBI). The project will provide better understanding of the patients' evolution during rehabilitation after TBI in terms of adaptation and social participation, assess the effect of rehabilitation and study social participation outcomes and quality of life of TBI patients one-year post-rehabilitation. Project benefits include improvement of clinical practices and support in decision-making.

The objectives of this research project are:

Part 1: To provide a picture of the evolution, in terms of social adaptation and participation of patients during rehabilitation after a TBI.

Part 2: To study social participation outcomes and quality of life of TBI individuals one year after the end of their rehabilitation.

DETAILED DESCRIPTION:
Context: This clinical research project is part of a series of innovative approaches to knowledge transfer in the field of trauma care funded by the Institut national d'excellence en santé et en services sociaux (INESSS) that have been recently conducted by 5 rehabilitation centers and which laid the groundwork for a culture of systematic measurement of clinical and functional evolution during rehabilitation and of social participation outcomes of Quebec adults with a traumatic brain injury (TBI). The Mayo-Portland Adaptability Inventory-4, or MPAI-4, which has three short scales: Abilities (12 items), Adaptation (12 items), Participation (8 items) giving specific indexes to each of these three dimensions, as well as a total score reflecting the general level of adaptation/social participation, was implemented in all the TBI rehabilitation programs within the trauma care continuum of greater Montreal (5 rehabilitation sites). These new practices allow to carry out original and rigorous prospective studies in order to better understand the multiple factors related to the clinical evolution of individuals who have sustained a TBI.

Objectives: Objective 1- To provide a picture of the evolution, in terms of social adaptation/participation, of a multicenter patient cohort in rehabilitation following TBI, according to their rehabilitation pathway (inpatient-outpatient, outpatient only); Objective Objective 2- To study social participation outcomes and quality of life of TBI individuals one year after the end of their rehabilitation.

Methodology: MPAI-4 data will be obtained for all patients at start and end of rehabilitation, and they will be subsequently contacted by phone one year after the end of their rehabilitation to administer the MPAI-4 Participation scale and QOLIBRI, measuring quality of life. At the end of the project, at least 1,500 unique patient cases will have been integrated into the study. For the one-year post-rehabilitation follow-up of the subjects included in the database we estimate the loss at 30% maximum; we expect to be able to collect post-rehabilitation data from a minimum of 700 patients who have completed rehabilitation. The raw data will be subjected to quantitative statistical analyzes to meet different objectives: ANOVAs to compare start-to-end rehabilitation measurement times for the different rehabilitation pathways; ANCOVA to compare groups on the total score and the three MPAI-4 scales at the end of rehabilitation, with scores at rehabilitation start as covariates; ANCOVA to compare the two groups on the Participation scale and QOLIBRI at the one-year follow-up with scores at rehabilitation start as covariates. Regression analyses will also be performed to determine which sociodemographic and clinical variables are most closely related to MPAI-4 and QOLIBRI scores.

Expected impacts: This innovative study will provide an unprecedented portrait of social participation and clinical evolution during rehabilitation within the continuum of trauma care services for a large cohort of adults (young adults, middle-aged adults, seniors) who sustained a TBI. This will provide evidence that will improve practices and support decision-making related to the organization of services. The systematic use of MPAI-4 may also help to assess the effects of changes in rehabilitation practices (eg, when implementing TBI practice guidelines). The various actors involved in this project and who will form the Monitoring committee will ensure the multiple benefits and impacts of the project.

ELIGIBILITY:
Inclusion Criteria:

* All adult TBI patients receiving post-acute rehabilitation services.

Exclusion Criteria:

* TBI patients that do not complete at least one month of rehabilitation.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a mild, moderate or severe TBI who are referred and registered in a multidisciplinary holistic rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from start of rehabilitation baseline (T0) Mayo-Portland Adaptability Inventory-4 (MPAI-4) at end of rehabilitation (post-intervention - T1) | Start to end of rehabilitation, an average of 1 year (pre-post rehabilitation - T0-T1)
  The MPAI-4 has 29 scored items and each item is scored on a 5-point scale (from 0 to 4). There are three subscales: Abilities (12 scored items, 0-47 after adjusting scores), Adjustment (9 scored items, 0-46 after adjusting scores), Participation (8 scored items, 0-30 after adjusting scores) giving specific indexes to each of these three dimensions, as well as a total score (all 29 items, 0-111) reflecting the general level of adaptation/social participation. As three items contribute to both the Adjustment and the Participation scales, the total score is less than the sum of the three subscales. Higher scores mean worse outcome.
Change from end of rehabilitation (T1) Mayo-Portland Adaptability Inventory-4 (MPAI-4) at 1-year post-rehabilitation (follow-up -T2) | 1 year post-rehabilitation (post-rehabilitation to 1-year follow-up - T1-T2)
  The MPAI-4 has 29 scored items and each item is scored on a 5-point scale (from 0 to 4). There are three subscales: Abilities (12 scored items, 0-47 after adjusting scores), Adjustment (9 scored items, 0-46 after adjusting scores), Participation (8 scored items, 0-30 after adjusting scores) giving specific indexes to each of these three dimensions, as well as a total score (all 29 items, 0-111) reflecting the general level of adaptation/social participation. As three items contribute to both the Adjustment and the Participation scales, the total score is less than the sum of the three subscales. Higher scores mean worse outcome.
Quality of Life after Brain Injury (QOLIBRI) status at 1-year post-rehabilitation | 1-year post-rehabilitation (T2)
  The MPAI-4 has 29 scored items and each item is scored on a 5-point scale (from 0 to 4). There are three subscales: Abilities (12 scored items, 0-47 after adjusting scores), Adjustment (9 scored items, 0-46 after adjusting scores), Participation (8 scored items, 0-30 after adjusting scores) giving specific indexes to each of these three dimensions, as well as a total score (all 29 items, 0-111) reflecting the general level of adaptation/social participation. As three items contribute to both the Adjustment and the Participation scales, the total score is less than the sum of the three subscales. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKerral, PhD, Principal Investigator — CRIR-IURDPM-CCSMTL and Université de Montréal
Locations (1):
- CRIR, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided